CLINICAL TRIAL: NCT02377843
Title: Making Effective HPV Vaccine Recommendations
Brief Title: Making Effective Human Papillomavirus (HPV) Vaccine Recommendations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other); North Carolina Department of Health and Human Services (Other Government); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 14-1873
Record Dates: First submitted 2015-02-27; First posted 2015-03-04 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: Human Papillomavirus
Keywords: vaccine; physician training; adolescent health
MeSH Terms: interventions — Community-Based Participatory Research

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Participatory (Experimental): This arm includes 10 pediatric or family medicine clinics located within a 2-hour driving distance of Chapel Hill, NC, and have 100 or more 11-12 year old patients with active records in the NCIR. Clinics randomized to the participatory study arm will receive a 1-hour in-person communication training.
  Interventions: Behavioral: Participatory
- Efficient (Experimental): This arm includes 10 pediatric or family medicine clinics located within a 2-hour driving distance of Chapel Hill, NC, and have 100 or more 11-12 year old patients with active records in the NCIR. Clinics randomized to the efficient study arm will receive a 1-hour in-person communication training.
  Interventions: Behavioral: Efficient
- Control (No Intervention): This arm includes 10 pediatric or family medicine clinics located within a 2-hour driving distance of Chapel Hill, NC, and have 100 or more 11-12 year old patients with active records in the NCIR. Clinics randomized to the control study arm will not receive a 1-hour in-person communication training.

INTERVENTIONS:
Behavioral: Participatory — The participatory intervention is a 1-hour training to help clinicians improve their ability to make strong and effective recommendations for HPV vaccine, and address parental concerns regarding HPV vaccination. The training includes four components:
  1. Review of information on HPV vaccine, including effectiveness, safety, rationale for targeting adolescents ages 11-12, and low HPV vaccine coverage rates compared to Tdap and meningococcal vaccine
  2. Skills building on how to recommend HPV vaccine using a participatory communication strategy based in shared decision making
  3. Practice using the communication strategy via role play
  4. Discussion on applying the communication strategy to medical practice
  Arms: Participatory
Behavioral: Efficient — The efficient intervention is a 1-hour training to help clinicians improve their ability to make strong and effective recommendations for HPV vaccine, and address parental concerns regarding HPV vaccination. The training includes four components:
  1. Review of information on HPV vaccine, including effectiveness, safety, rationale for targeting adolescents ages 11-12, and low HPV vaccine coverage rates compared to Tdap and meningococcal vaccine
  2. Skills building on how to recommend HPV vaccine using an efficient communication strategy based on first announcing the child is due for 3 vaccines
  3. Practice using the communication strategy via role play
  4. Discussion on applying the communication strategy to medical practice
  Arms: Efficient

SUMMARY:
Coverage of HPV vaccination among US teens is low, far below Healthy People 2020 goals. A central reason for low coverage is infrequent and inadequate healthcare provider recommendation of HPV vaccine. The proposed intervention aims to train clinicians to provide effective recommendations for the vaccine using participatory or efficient communication strategies.

This study will evaluate the effectiveness of two communication trainings to increase HPV vaccination coverage among adolescent patients. We will compare HPV vaccination for pediatric and family medicine clinics receiving a participatory communication training, efficient communication training, or no training. Ten clinics will be randomly assigned to each study arm for a total of 30 clinics. The primary outcome of this study is to compare the change in clinics' levels of HPV vaccination initiation coverage among 11-12 year old adolescent patients from baseline to 6 month follow-up. Secondarily, we will compare the change in HPV vaccination initiation coverage in 13-17 year old adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Eligible clinics are pediatric and family medicine practice clinics located within a 2-hour driving distance of Chapel Hill, NC, and have 100 or more 11-12 year old patients with active records in the NCIR. Clinics must have at least one pediatric or family medicine physician who provides HPV vaccine to adolescents ages 11-12.

Exclusion Criteria:

* Ineligible clinics include those that have participated in a quality improvement study to increase HPV vaccination rates in the last 6 months or plan to participate in such a study in the next 6 months.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
6 month % change in HPV vaccination (≥ 1 dose), control vs. each intervention arm (efficient or participatory), 11-12 year olds | Baseline, month 6
  Analysis controlling for sex. Vaccination as measured by North Carolina Immunization Registry (NCIR).

SECONDARY OUTCOMES:
6 month % change in HPV vaccination (≥ 1 dose), efficient arm vs. participatory arm, 11-12 year olds | Baseline, month 6
  Analysis controlling for sex. Vaccination as measured by NCIR.
3 month % change in HPV vaccination (≥ 1 dose), control vs. each intervention arm, 11-12 year olds | Baseline, month 3
  Analysis controlling for sex. Vaccination as measured by NCIR.
3 month % change in HPV vaccine completion (3 doses), control vs. each intervention arm, 11-12 year olds | Baseline, month 3
  Analysis controlling for sex. Vaccination as measured by NCIR.
6 month % change in HPV vaccine completion (3 doses), control vs. each intervention arm, 11-12 year olds | Baseline, month 6
  Analysis controlling for sex. Vaccination as measured by NCIR.
3 month % change in tetanus, diphtheria, and acellular pertussis (Tdap) vaccination, control arm vs. each intervention arm, 11-12 year olds | Baseline, month 3
  Vaccination as measured by NCIR.
6 month % change in Tdap vaccination, control arm vs. each intervention arm, 11-12 year olds | Baseline, month 6
  Vaccination as measured by NCIR.
3 month % change in meningococcal vaccination (≥ 1 dose), control arm vs. each intervention arm, 11-12 year olds | Baseline, month 3
  Vaccination as measured by NCIR.
6 month % change in meningococcal vaccination (≥ 1 dose), control arm vs. each intervention arm, 11-12 year olds | Baseline, month 6
  Vaccination as measured by NCIR.
3 month % change in HPV vaccination (≥ 1 dose), control vs. each intervention arm, 13-17 year olds | Baseline, month 3
  Analysis controlling for sex. Vaccination as measured by NCIR.
6 month % change in HPV vaccination (≥ 1 dose), control vs. each intervention arm, 13-17 year olds | Baseline, month 6
  Analysis controlling for sex. Vaccination as measured by NCIR.
3 month % change in HPV vaccine completion (3 doses), control vs. each intervention arm, 13-17 year olds | Baseline, month 3
  Analysis controlling for sex. Vaccination as measured by NCIR.
6 month % change in HPV vaccine completion (3 doses), control vs. each intervention arm, 13-17 year olds | Baseline, month 6
  Analysis controlling for sex. Vaccination as measured by NCIR.
3 month % change in Tdap vaccination, control arm vs. each intervention arm, 13-17 year olds | Baseline, month 3
  Vaccination as measured by NCIR.
6 month % change in Tdap vaccination, control arm vs. each intervention arm, 13-17 year olds | Baseline, month 6
  Vaccination as measured by NCIR.
3 month % change in meningococcal vaccination (≥ 1 dose), control arm vs. each intervention arm, 13-17 year olds | Baseline, month 3
  Vaccination as measured by NCIR.
6 month % change in meningococcal vaccination (≥ 1 dose), control arm vs. each intervention arm, 13-17 year olds | Baseline, month 6
  Vaccination as measured by NCIR.
Change in clinician HPV vaccine knowledge, efficient arm vs. participatory arm | Pre-training, Post-training
  3-item knowledge scale (low vaccine coverage, vaccine effectiveness, recommendation impact on vaccine uptake).
Change in clinician self-efficacy, efficient arm vs. participatory arm | Pre-training, Post-training, week 2
  2-item self-efficacy scale (effectively recommending HPV vaccination, addressing parents' concerns).
Change in clinician recommendation quality, efficient arm vs. participatory arm | Pre-training, week 2
  4-item recommendation quality scale (urgency, consistency, timeliness, strength of endorsement) (Gilkey et al.).
Change in clinician communication of routine use, efficient arm vs. participatory arm | Pre-training, Post-training, week 2
  1 item on communicating HPV vaccination as part of routine adolescent care.
Change in clinician communication of HPV vaccination as cancer prevention, efficient arm vs. participatory | Pre-training, Post-training, week 2
  1 item on communicating HPV vaccination as cancer prevention.
3 month % change in HPV vaccination (≥ 1 dose), control vs. each intervention arm, 11-12 year old females | Baseline, month 3
  Vaccination as measured by NCIR.
3 month % change in HPV vaccination (≥ 1 dose), control vs. each intervention arm, 11-12 year old males | Baseline, month 3
  Vaccination as measured by NCIR.
6 month % change in HPV vaccination (≥ 1 dose), control vs. each intervention arm, 11-12 year old females | Baseline, month 6
  Vaccination as measured by NCIR.
6 month % change in HPV vaccination (≥ 1 dose), control vs. each intervention arm, 11-12 year old males | Baseline, month 6
  Vaccination as measured by NCIR.
3 month % change in HPV vaccine completion (3 doses), control vs. each intervention arm, 11-12 year old females | Baseline, month 3
  Vaccination as measured by NCIR.
3 month % change in HPV vaccine completion (3 doses), control vs. each intervention arm, 11-12 year old males | Baseline, month 3
  Vaccination as measured by NCIR.
6 month % change in HPV vaccine completion (3 doses), control vs. each intervention arm, 11-12 year old females | Baseline, month 6
  Vaccination as measured by NCIR.
6 month % change in HPV vaccine completion (3 doses), control vs. each intervention arm, 11-12 year old males | Baseline, month 6
  Vaccination as measured by NCIR.
3 month % change in HPV vaccination (≥ 1 dose), control vs. each intervention arm, 13-17 year old females | Baseline, month 3
  Vaccination as measured by NCIR.
3 month % change in HPV vaccination (≥ 1 dose), control vs. each intervention arm, 13-17 year old males | Baseline, month 3
  Vaccination as measured by NCIR.
6 month % change in HPV vaccination (≥ 1 dose), control vs. each intervention arm, 13-17 year old females | Baseline, month 6
  Vaccination as measured by NCIR.
6 month % change in HPV vaccination (≥ 1 dose), control vs. each intervention arm, 13-17 year old males | Baseline, month 6
  Vaccination as measured by NCIR.
3 month % change in HPV vaccine completion (3 doses), control vs. each intervention arm, 13-17 year old females | Baseline, month 3
  Vaccination as measured by NCIR.
3 month % change in HPV vaccine completion (3 doses), control vs. each intervention arm, 13-17 year old males | Baseline, month 3
  Vaccination as measured by NCIR.
6 month % change in HPV vaccine completion (3 doses), control vs. each intervention arm, 13-17 year old females | Baseline, month 6
  Vaccination as measured by NCIR.
6 month % change in HPV vaccine completion (3 doses), control vs. each intervention arm, 13-17 year old males | Baseline, month 6
  Vaccination as measured by NCIR.

CONTACTS AND LOCATIONS:
Overall Officials: Noel T Brewer, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Melissa B Gilkey, PhD, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (1):
- University of North Carolina, Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Malo TL, Hall ME, Brewer NT, Lathren CR, Gilkey MB. Why is announcement training more effective than conversation training for introducing HPV vaccination? A theory-based investigation. Implement Sci. 2018 Apr 19;13(1):57. doi: 10.1186/s13012-018-0743-8. PMID 29673374
- [Derived] Brewer NT, Hall ME, Malo TL, Gilkey MB, Quinn B, Lathren C. Announcements Versus Conversations to Improve HPV Vaccination Coverage: A Randomized Trial. Pediatrics. 2017 Jan;139(1):e20161764. doi: 10.1542/peds.2016-1764. Epub 2016 Dec 5. PMID 27940512